CLINICAL TRIAL: NCT01962831
Title: Randomized Controlled Trial: Single Balloon Catheter Versus Dinoprostone Vaginal Insert for Induction of Labour of Women With a BMI Equal to or Greater Than 30
Brief Title: Randomized Controlled Trial: Induction of Labour of Obese Women With Dinoprostone or Single Balloon Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saskatchewan Health Authority - Regina Area (Other)
Responsible Party: Principal Investigator, Dr. Christine Lett, Clinical Assistant Professor of Obstetrics & Gynecology, University of Saskatchewan, Saskatchewan Health Authority - Regina Area
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB-13-51
Record Dates: First submitted 2013-09-19; First posted 2013-10-14 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Obesity; Pregnancy; Labor, Induced
Keywords: obesity; labor, induced; pregnancy; cervical ripening; dinoprostone
MeSH Terms: conditions — Obesity | interventions — Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dinoprostone (Experimental): Group of women that will receive dinoprostone for induction of labour dinoprostone 10 mg in vagina to be reassessed every 24 hours
  Interventions: Drug: Dinoprostone
- Single balloon foley catheter (Experimental): Group of women that will have a single balloon foley catheter inserted for induction of labour
  Interventions: Device: Single balloon foley catheter

INTERVENTIONS:
Drug: Dinoprostone
  Other Names: Cervidil
  Arms: dinoprostone
Device: Single balloon foley catheter
  Arms: Single balloon foley catheter

SUMMARY:
The purpose of this study is to compare the efficacy of single balloon foley catheters to dinoprostone for the induction of labour of obese women. The investigators suspect that women assigned to the foley group will have a shorter induction to delivery time than women in the dinoprostone group.

ELIGIBILITY:
Inclusion Criteria:

* Obese (BMI >30 before 20 weeks gestational age)
* Singleton pregnancy
* Vertex presentation
* Bishop Score <6
* Intact membranes
* Gestational age 37+0 to 42+0
* Normal fetal heart tracing on admission for ripening

Exclusion Criteria:

* Induction of labour for intrauterine fetal demise
* Intrauterine growth restriction
* Suspected abruption at the start of induction
* Any contraindication for a vaginal delivery

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Time(hours) from initiation of induction of labour to vaginal delivery | Will be assessed at the end of each vaginal delivery

SECONDARY OUTCOMES:
Number of vaginal deliveries within 24 hours in each group | 2 years
Number of cesarean sections in each group | 2 years
Number of operative vaginal deliveries in each group | 2 years
Number of chorioamnionitis cases in each group | 2 years
Number of patients that required oxytocin administration in each group | 2 years
Number of patients that required an epidural in each group | 2 years
Number of babies that required neonatal intensive care unit (NICU) admission in each group | 2 years
Number of babies that had an arterial pH <7 in each group | 2 years
Number of babies that had an APGAR score <7 at 5 minutes | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Christine Lett, MD, Principal Investigator — Saskatchewan Health Authority - Regina Area
Locations (1):
- Regina Qu'Appelle Health Region, Regina, Saskatchewan, Canada